CLINICAL TRIAL: NCT03151902
Title: Detection of Viral Particels in Urticaria Patients
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Menachem Rottem, Head, Allergy Asthma and Immunology, HaEmek Medical Center, Israel
Other Study IDs: HaEmekMC1
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Urticaria Chronic
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blood samples from urticaria patients will be analyzed for viral particles

DETAILED DESCRIPTION:
After digestion with DNase to eliminate human DNA, RNA will be reversed-transcribed and amplified with random primer/ Amplification products will be pooled and sequenced/ After substruction of sequences of vertebrates and highly repetitive sequences, contiguous sequences will be assembled and compared with motifs represented in databases of viruses. which will enable identification of putative protein sequences consistent with viruses

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic spontaneous urticaria

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic spontaneous urticaria
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-07-02 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
viral particles | 6 months
  presence of viral particels

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Rottem, Principal Investigator — haemek medical center
Locations (1):
- Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No